CLINICAL TRIAL: NCT00934440
Title: A Phase I/II Study Evaluating The Efficacy OF 5-Azacitidine And Bevacizumab In Advanced Renal Cell Carcinoma
Brief Title: A Study to Evaluate the Effectiveness of 5-Azacitidine and Bevacizumab in Advanced Renal Cell Carcinoma
Acronym: 5-AZ
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11570
Record Dates: First submitted 2009-06-23; First posted 2009-07-08 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Renal Cell Carcinoma
Keywords: kidney cancer; renal cell
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bevacizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation: 5-azacitidine (Experimental): A traditional 3+3 dose escalation trial was implemented. Successive cohorts of patients (3 participants/cohort) received bevacizumab at the standard dose of 10mg/kg in combination with escalating doses of 5-azacitidine. If no dose limiting toxicity (DLT) is seen, subsequent patients will be treated at the next dose level. If one DLT is seen, an additional three patients will be accrued at that dose level. If two or more DLTs are seen at one dose level, then the previous dose level will be chosen for phase IIA. If two DLT's are seen at dose level 1, the trial will end. The standard 5-azacitidine dose is 75mg/m2/day for 7 days. If no DLT is seen at dose level 3, then we will proceed with the phase IIA portion of the study.
  Interventions: Drug: Bevacizumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Bevacizumab — * First treatment: 10 milligram per kilograms (MG/KG) intravenously (IV) on Day 1every two weeks over 90 minutes.
  * Second treatment: 10 MG/KG IV on Day 1 every two weeks over 60 minutes.
  * Third and subsequent treatments: 10 MG/KG IV on Day 1 every two weeks over 30 minutes (minimum of two cycles).
  Other Names: Avastin
Drug: Azacitidine — * Dose level 1: 35 mg/m2/day for 7 days.
  * Dose level 2: 55 mg/m2/day for 7 days.
  * Dose level 3: 75 mg/m2/day for 7 days.
    * mg/m2/day = dose based on height and weight
  Other Names: Vidaza

SUMMARY:
To identify the maximum tolerable dose and assess qualitative/quantitative toxicities in patients with advanced renal cell cancer treated with combination of 5-azacitidine and bevacizumab.

DETAILED DESCRIPTION:
In this study, the investigator will assess progression-free and overall survival of patients with advanced renal cell carcinoma treated with 5-azacitidine in combination with bevacizumab. Patients will continue on treatment until either disease progression or development of other criteria for withdrawal.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years old
* ECOG Performance Status 0, 1 or 2
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count(ANC)>1,500/mm3
  * Platelet count >100,000/mm3
  * Total bilirubin < 1.5 times ULN
  * ALT and AST < 2.5 times the ULN (< 5 x ULN for patients with liver involvement)
  * Creatinine < 1.5 times ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for duration of study. Men should use adequate birth control for at least 3 months after the last administration of Bevacizumab.
* Ability to understand and willingness to sign written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Patients not on anticoagulation must have an INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of treatment and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Must have histologically or cytologically confirmed renal cell carcinoma which is metastatic (M1). Patients with unresectable primary tumors (but MO) are eligible.
* Must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension. Soft tissue disease that has been radiated in the 2 months prior to registration is not assessable as measurable disease. Soft tissue disease within a prior radiation field must have progressed to be considered assessable. X-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration. X-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration.
* Patients with metastatic disease who have a resectable primary tumor and deemed a surgical candidate may have undergone resection and have recovered from surgery. At least 28 days must have elapsed since surgery and must have recovered from any adverse effects of surgery.
* Urine protein must be screened by urine analysis for Urine Protein Creatinine (UPC) ratio. For UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1,000mg for patient enrollment. The urine protein used to calculate the UPC ratio must be obtained within 28 days prior to registration. NOTE: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1gm. UPC ratio is calculated using one of the following formulas: [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL
* May have received prior immunotherapy with either interferon (IFN) and/or Interleukin-2 (IL-2) or the combination of IFN/IL2 or prior chemotherapy (ie, gemcitabine and capecitabine).
* Must have failed at least 1 prior biologic agent (sunitinib, sorafenib, or temsorlimus). No limit on the number of prior therapies.
* At least 14 days must have elapsed since the last treatment. Must have recovered from any adverse effects of prior therapy.
* May have received prior radiation therapy. At least 21 days must have elapsed since completion of prior radiation therapy. Must have recovered from all associated toxicities at the time of registration.
* Pregnant or nursing women not eligible because of potential teratogenic side effects of 5-azacitidine and bevacizumab on the developing fetus or nursing infant. Women and men of reproductive potential must have agreed to use an effective contraceptive method.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-azacitidine or bevacizumab are not eligible.
* Involvement in correlative studies must be offered to all patients but is not required.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which patient is currently in complete remission, or any other cancer from which patient has been disease-free for 2 years.
* Must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria

* Cardiac disease: Congestive heart failure > class II NYHA. Must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of brain to exclude brain metastasis.
* Patients who have received prior bevacizumab are eligible for phase I portion of study but ineligible for phase II study.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombosis or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months. Patients with tumor related IVC thrombosis are eligible.
* Serious non-healing wound, ulcer, or bone fracture.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Van Veldhuizen, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Stormont-Vail Cotton O'Neil Cancer Center, Topeka, Kansas

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I 5-Azacitidine Maximum Tolerated Dose (MTD): All patients in phase I and II will receive bevacizumab at the standard dose of 10mg/kg IV every two weeks. The first dose should be infused over 90 minutes. If no adverse reactions occur, the second dose of bevacizumab should be given over a minimum of 60 minutes. If no adverse event occurs, third and subsequent doses should be administered over a minimum of 30 minutes.
Period: Overall Study
Arm/Group | Phase I 5-Azacitidine Maximum Tolerated Dose (MTD)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase I 5-Azacitidine Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Toxicities by Dose Level
Description: Toxicities determined using Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: 3 to 6 months
Measure: Number; unit: adverse events
Arm/Group | 5-Azacitidine Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 11
adverse events
  AEs at dose level 1 | 44
  AEs at dose level 2 | 48
  AEs at dose level 3 | 49

2. Secondary Outcome: Time to Progression
Description: The time to progression was measured using time from the first day of treatment to the first day of an evaluation of progressive disease or the date of death for any cause.
Time Frame: 2 years
Measure: Mean (Full Range); unit: months
Groups:
- Dose Escalation: 5-azacitidine: A traditional 3+3 dose escalation trial was implemented. Successive cohorts of patients (3 participants/cohort) received bevacizumab at the standard dose of 10mg/kg in combination with escalating doses of 5-azacitidine. If no dose limiting toxicity (DLT) is seen, subsequent patients will be treated at the next dose level. If one DLT is seen, an additional three patients will be accrued at that dose level. If two or more DLTs are seen at one dose level, then the previous dose level will be chosen for phase IIA. If two DLT's are seen at dose level 1, the trial will end. The standard 5-azacitidine dose is 75mg/m2/day for 7 days. If no DLT is seen at dose level 3, then we will proceed with the phase IIA portion of the study.
  Bevacizumab:
  * First treatment: 10 milligram per kilograms (MG/KG) intravenously (IV) on Day 1
  * Second treatment: 10 MG/KG IV on Day 1
  * Third and subsequent treatments: 10 MG/KG IV on Day 1
Arm/Group | Dose Escalation: 5-azacitidine
Number analyzed (Participants) | 11
months | 5.6 [1.0 to 22.8]

ADVERSE EVENTS:
Time Frame: 2 years, 1 month
Arm/Group | Phase I 5-Azacitidine Maximum Tolerated Dose (MTD)
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I 5-Azacitidine Maximum Tolerated Dose (MTD) (N=11)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I 5-Azacitidine Maximum Tolerated Dose (MTD) (N=11)
Abdominal pain (Gastrointestinal disorders) | 3
Adrenal insufficiency (Endocrine disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 — elevated ABG
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dyspnea (Ear and labyrinth disorders) | 4
Edema limbs (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Infection (Infections and infestations) | 1 — Influenza A
Injection site reaction (Skin and subcutaneous tissue disorders) | 6
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 1
D-dimer 1837 (Metabolism and nutrition disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neutrophils (Blood and lymphatic system disorders) | 2
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
tachypnea (Respiratory, thoracic and mediastinal disorders) | 1
rales (scattered) (Respiratory, thoracic and mediastinal disorders) | 1
rhonchi (scattered) (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Taste alteration (Gastrointestinal disorders) | 1
Thrombosis/embolism (vascular access) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight gain (General disorders) | 1
Weight loss (General disorders) | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes